CLINICAL TRIAL: NCT07237997
Title: Re-examining Nutrition in Dialysis Patients: Nutritional Losses and the Role of Supplementation (Part 2).
Brief Title: Protein Supplementation During Dialysis (PROSED)
Acronym: PROSED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25032; SG_AHPF_001_20221129 (Other Grant/Funding Number: Kidney Research UK)
Record Dates: First submitted 2025-07-18; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Dialysis Patients; Dialysis; Protein Energy Wasting; Protein Intake; High Protein Dietary Intake; Diet; Diet Therapy; Hospitalisation; Muscle Mass and Strength; Muscle Mass

STUDY DESIGN:
Intervention Model Description: This is an interventional pilot study of protein supplementation to test the hypothesis that a higher dietary protein intake is associated with a reduced unplanned hospitalisation admission rate over 2 years.
  The investigators will aim to recruit 114 participants with randomisation stratified across dialysis modalities (ICHD, CAPD, APD, HHD, NHD). Recruitment proportions will align with current dialysis populations at the study units - i.e., approximately 10-15% CAPD, 10-15% APD, 5-10% HHD, 3-5% NHD and 60-70% ICHD.
  Description of the intervention Once consented, participants will be randomly assigned to a high-protein group or usual care.
  Higher and usual protein intake targets, referred as individualised protein supplementation regimen, will be set within the limits of previously published mortality data Higher protein intake will aim to achieve 1.4g protein per kg of dry body weight per day usual protein intake will aim to achieve at least 1.0g protein per kg of dry body weight
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Protein Arm (No Intervention): In the Standard Protein Arm, participants will aim to consume at least 1.0g of protein per kg of dry body weight.
- High Protein Arm (Experimental): In the High Protein arm, participants will need to consume 1.4g of protein per kg of dry body weight a day and protein supplements will be used to achieve this (Renapro and Renapro shot)
  Interventions: Dietary Supplement: High Protein Diet/Modular protein supplements will be used

INTERVENTIONS:
Dietary Supplement: High Protein Diet/Modular protein supplements will be used — High Protein Diet/Supplements 1.4g/kg/body weight/day
  Arms: High Protein Arm

SUMMARY:
When a patient has dialysis some nutrients are lost in the process. Nutritional losses include protein, trace elements (i.e. zinc, copper and selenium) and water-soluble vitamins (Vitamins C and B). These nutrients are essential for normal body function, including a good immune system and nutritional status. For example, on average the protein losses during a dialysis session (the process where the blood is cleaned via a machine and special fluid) is equal to 6g of protein/day (which is the equivalent of the amount of protein in 1 egg). Protein needs for the general population are 0.8g protein per kg of body weight. Because people on dialysis lose protein via the dialysis, it is thought that these people need to eat more protein. Currently, in clinical practice for people receiving dialysis, the guidelines are to aim for 1.1 -1.4g of protein per kg of body weight. However, the research is old and very weak.

Dialysis treatments have changed over the past 40 years, and the investigator does not know if the replacement of these nutritional losses is important to how well people do on dialysis and if they have any effect on survival. Previous research is mostly limited to haemodialysis (a type of dialysis that requires a machine which cleans the patients' blood via special filters) and peritoneal dialysis (this is a type of dialysis which happens via the patients' tummy). There is no research on the nutritional supplementation in home HD and nocturnal HD. Our research will investigate if a higher protein provision leads to a reduction is hospital admissions and improved outcomes in patients receiving dialysis.

DETAILED DESCRIPTION:
Malnutrition, specifically protein-energy wasting (PEW), is a major independent risk factor for poor quality of life and premature death in patients receiving dialysis.

Nutritional losses occur in patients on dialysis and have been documented over 40 years . Nutritional losses include nitrogen (amino acids, small peptides, proteins), trace elements (i.e. zinc, copper and selenium) and water-soluble vitamins (i.e. B vitamins and vitamin C). Dialysis membranes and modalities have changed over the past 40 years, and the investigators do not know if these nutritional losses (and their replacement) are of clinical significance to patients' clinical outcomes. In addition, research on this topic has focused on in-centre haemodialysis (ICHD), and, to a lesser extent, on peritoneal dialysis (PD). There are no studies reporting nutritional losses in patients receiving HD at home (HHD) and nocturnal HD (NHD) where different technologies and scheduling are often utilised. Nutritional losses could be different for different dialysis modalities. While there has been a lot of observational cohort data looking at different levels of protein intake, no long-term interventional studies have been conducted.

Funding was successfully obtained by Kidney Research UK to conduct two studies:

* Phase one, which is currently ongoing (IRAS 320440), aims to measure nutritional losses in people receiving maintenance dialysis, in different dialysis modalities.
* Phase two, this study (IRAS 343782), is a pragmatic pilot interventional study which will assess the impact of different protein intakes on patients' clinical outcomes in people on maintenance dialysis.

Dialysis techniques and modalities have changed significantly over the past 20 years. Yet current guidelines for protein provision are based on out-of-date data. Clinical guidelines for protein provision in ICHD and PD have not changed significantly in the past 20 years. There are no guidelines for HHD and NHD, as there is no evidence.

There are no main ethical or legal issues associated with this study. The primary aim of the study is to assess the association between hospitalisation rate and protein intake over a 2-year period.

Secondary objectives include associations between protein intake and mortality, cardiovascular outcomes, biophysical parameters, medication usage (such as erythropoietin, antibiotics, as well as other medication), infection rates, nutritional status (including anthropometry, body composition and functional markers of muscle mass) and quality of life indices

This study will be part two of a feasibility study where the investigators will assess whether protein supplementation impacts patient clinical outcomes. In part one, the investigators evaluated the protein losses in different dialysis modalities and measured nitrogen balance with stable isotopes (IRAS 320440).

The investigators know that there are protein losses via haemodialysis, peritoneal dialysis, home haemodialysis and nocturnal haemodialysis.

Participants will have a detailed nutritional assessment (including measurement of body composition), and their protein intake will be estimated at regular intervals for 2 years.

There are logistical issues in measuring nutritional status at each patient's home and these will be addressed by liaising with the home therapy team and coinciding nutritional assessment with patients' hospital visit as part of their standard care. Furthermore, patients will be asked to collect 24-hour urine collections (if they pass urine) at regular intervals. No additional blood samples will be needed (in addition to those required for standard care). These issues were discussed with our local team as well as by the patient representative group from Kidney Research UK, who acknowledged that this study is unlikely to carry a significant burden to participants.

There is no conflict of interest with this study.

Our research will fully engage with our patient and public involvement (PPI) group at the time of study design, during the research and upon completion. The investigators intend to schedule sample acquisition and study visits around standard therapies to minimise requirements for additional site visits. PPI input will be sought to confirm how the trial design can be optimised to minimise inconvenience to patients and maximise recruitment.

At the end of study, all participants will be informed of the overall findings with a written report in lay language, easy to understand.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (no upper age limit)
* Patients receiving maintenance dialysis for ≥ three months
* Ability to provide informed consent

Exclusion Criteria:

* Anticipated live donor kidney transplant and/or kidney recovery within the period of sample collection.
* Anticipated change of dialysis modality within the period of sample collection
* Severe malnutrition based on either:

  * Renal 7-point Subjective Global Assessment (SGA) scores of 1-2
  * Global Leadership Initiative Malnutrition (GLIM) Stage 2
* Protein-losing enteropathy.
* Persistent nephrotic syndrome with >3g/day urinary protein loss.
* Active wounds or burns contributing to protein losses as judged by the investigator.
* Current active acute inflammatory illness (likely to have catabolic effect in the opinion of the investigator).
* Current malignancy based on recent (<12 months) diagnosis and/or active treatment for malignancy and/or planned treatment for malignancy, excluding non-melanoma skin cancers.
* Pregnancy (current or planned within duration of study) or breast feeding.
* People with swallowing difficulties precluding safe ingestion (International Dysphagia Diet Standardization Initiative (IDDSI) level 0 thin fluid).
* People receiving intradialytic parenteral nutrition or intra-peritoneal amino acids, or any other forms of artificial feeding
* People prescribed levodopa
* People who are receiving chronic glucocorticoid therapy (>10mg day prednisolone or equivalent for >7 days within preceding 90 days).
* People who are consuming a protein dietary intake above 1.5g protein/kg/body weight.
* People who, in the opinion of the investigator, will be unable to comply with study protocol requirements.
* People who are vegan or other religious based dietary restrictions which would prevent them taking the supplement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
To identify how protein intake and supplements influence patients' unplanned hospitalisation rate. | 2 years
  Purpose
  To measure the impact of different amounts of protein intake (protein in the diet) on clinical outcomes (including unplanned hospital admissions) in patients receiving the different dialysis modalities (ICHD, HHD, NHD and PD).
  The investigators hypothesis is that a modality-specific and high-protein supplementation regimen reduces unplanned hospitalisation rate in patients receiving dialysis (ICHD, PD, HD, NHD) compared with those without supplementation.

SECONDARY OUTCOMES:
To assess association between protein intake and patients related outcomes measures. | 2 years
  To assess the correlation between protein intake and:
  * the rate of mortality
  * the incidence of cardiovascular events
  * % of patients of specific medications (such as erythropoietin, antibiotics, as well as other medications)
  * infection rates
  * nutritional status , including body composition (measured via bioimpedence in kg of fat mass and kg fat free mass, calf circumference in cm), functional markers of muscle mass (measured via hand grip strength in kg and hand grip index)
  * quality of life will be measure via a scales SF-36 and EuroQoL-5D
  The following assessments will be performed using the following measurements:
  Chronic Kidney Disease physical activity questionnaire Karnofsky score Subjective Global Assessment Global Leadership Initiative malnutrition tool Clinical Frailty score Malnutrition Inflammation score Sarcopenia -F tool

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Selby, BMedSci BMBS DM, Principal Investigator — University of Nottingham
Locations (1):
- Centre for Kidney Research and Innovation (CKRI), Academic Unit for Translational Medical Sciences School of Medicine (Royal Derby Hospital Campus), Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
If there is a need to share the IPD based on the findings of this study, a table will be included with the relevant data

REFERENCES:
- [Background] Sahathevan S, Khor BH, Ng HM, Gafor AHA, Mat Daud ZA, Mafra D, Karupaiah T. Understanding Development of Malnutrition in Hemodialysis Patients: A Narrative Review. Nutrients. 2020 Oct 15;12(10):3147. doi: 10.3390/nu12103147. PMID 33076282
- [Background] Zazzeroni L, Pasquinelli G, Nanni E, Cremonini V, Rubbi I. Comparison of Quality of Life in Patients Undergoing Hemodialysis and Peritoneal Dialysis: a Systematic Review and Meta-Analysis. Kidney Blood Press Res. 2017;42(4):717-727. doi: 10.1159/000484115. Epub 2017 Oct 19. PMID 29049991
- [Background] Mafrici B, Armstrong-Brown V. Protein-energy wasting and nutritional requirements in dialysis. Journal Kidney Care 2017 2 (2), https://doi.org/10.12968/jokc.2017.2.2.
- [Background] Hanna RM, Ghobry L, Wassef O, Rhee CM, Kalantar-Zadeh K. A Practical Approach to Nutrition, Protein-Energy Wasting, Sarcopenia, and Cachexia in Patients with Chronic Kidney Disease. Blood Purif. 2020;49(1-2):202-211. doi: 10.1159/000504240. Epub 2019 Dec 18. PMID 31851983
- [Background] Viramontes-Horner D, Pittman Z, Selby NM, Taal MW. Impact of malnutrition on health-related quality of life in persons receiving dialysis: a prospective study. Br J Nutr. 2022 Jun 14;127(11):1647-1655. doi: 10.1017/S000711452100249X. Epub 2021 Jul 5. PMID 34218825
- [Background] Kittiskulnam P, Chuengsaman P, Kanjanabuch T, Katesomboon S, Tungsanga S, Tiskajornsiri K, Praditpornsilpa K, Eiam-Ong S. Protein-Energy Wasting and Mortality Risk Prediction Among Peritoneal Dialysis Patients. J Ren Nutr. 2021 Nov;31(6):679-686. doi: 10.1053/j.jrn.2020.11.007. Epub 2021 Feb 25. PMID 33642190
- [Background] Sabatino A, Regolisti G, Karupaiah T, Sahathevan S, Sadu Singh BK, Khor BH, Salhab N, Karavetian M, Cupisti A, Fiaccadori E. Protein-energy wasting and nutritional supplementation in patients with end-stage renal disease on hemodialysis. Clin Nutr. 2017 Jun;36(3):663-671. doi: 10.1016/j.clnu.2016.06.007. Epub 2016 Jun 18. PMID 27371993
- See also: Lay Summary of Research Project from Kidney Research UK: What is the impact of different types of dialysis on levels of protein? — https://www.kidneyresearchuk.org/2023/08/03/what-is-the-impact-of-different-types-of-dialysis-on-levels-of-protein/